CLINICAL TRIAL: NCT00112892
Title: A Phase I and Pharmacokinetic Study of Selenomethionine With Fixed Dose Irinotecan in Advanced Solid Tumors
Brief Title: Irinotecan and Selenium in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000427616; RPCI-I-32804
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Selenium; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: selenium
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Selenium may allow higher doses of irinotecan to be given. Giving irinotecan together with selenium may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of selenium when given together with irinotecan in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the optimal loading and maintenance doses of selenium necessary to achieve selenium concentrations exceeding 15 μM when administered with irinotecan in patients with advanced solid tumors.

Secondary

* Determine the pharmacokinetics of this regimen in these patients.
* Determine the toxic effects of this regimen in these patients.
* Determine any observed tumor response to this regimen in these patients.

OUTLINE: This is a dose-escalation study of selenium.

Patients receive a loading dose* of oral selenium twice daily on days -6 to 0. Patients then receive oral selenium once daily on days 1-42 and irinotecan IV over 90 minutes on days 1, 8, 15, and 22. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

NOTE: *The loading dose is administered prior to course 1 only.

Cohorts of 3-6 patients receive escalating doses of selenium until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 2-36 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Metastatic or unresectable disease
* Standard curative or palliative treatments do not exist or are no longer effective OR treatment with single-agent irinotecan does not constitute a reasonable treatment option
* No known untreated or progressive brain metastases

  * Previously treated brain metastases allowed provided all of the following are true:

    * No significant neurological deficit
    * No requirement for anti-epileptic medications
    * Disease stable by brain CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 12 weeks

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT ≤ 3 times upper limit of normal
* Albumin ≥ 3.0 g/dL
* No Gilbert's disease

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No clinically significant cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to receive oral medications
* No active inflammatory bowel disease or chronic diarrhea
* No known HIV positivity
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study drugs
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for carmustine or mitomycin)

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2004-08; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Fakih MG, Pendyala L, Brady W, Smith PF, Ross ME, Creaven PJ, Badmaev V, Prey JD, Rustum YM. A Phase I and pharmacokinetic study of selenomethionine in combination with a fixed dose of irinotecan in solid tumors. Cancer Chemother Pharmacol. 2008 Aug;62(3):499-508. doi: 10.1007/s00280-007-0631-4. Epub 2007 Nov 8. PMID 17989978